CLINICAL TRIAL: NCT05110729
Title: Quality of Life and Life Satisfaction in Pediatric and Adolescent Gymnasts Through Injury
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-4271
Record Dates: First submitted 2021-10-22; First posted 2021-11-08 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Injury; Quality of Life
Keywords: Gymnastics; Quality of Life and Life Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study aims to assess the quality and life and life satisfaction of pediatric and adolescent gymnasts throughout their musculoskeletal injury recovery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female gymnasts ages 8-18 years old
* Participating in Excel or Developmental gymnastics programs who present to Children's Hospital Colorado sports medicine or orthopedic clinics with a musculoskeletal injury.

Exclusion Criteria:

* Gymnasts only participating in Colorado Association for Recreational Athletics (CARA) gymnastics, retired gymnasts, and adult or collegiate gymnasts.
* Vulnerable populations (prisoners, pregnant women, individuals with decreased decision making capacity(

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from Children's Hospital Colorado Sports medicine and Orthopedic outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1218 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | 1 day Initial Visit
  A validated questionnaire that quantifies quality of life and life satisfaction in pediatric and adolescent populations.
Patient-Reported Outcomes Measurement Information System (PROMIS) | At follow up visit, up to 3 months post initial visit
  A validated questionnaire that quantifies quality of life and life satisfaction in pediatric and adolescent populations.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 1 day (At clearance visit to return to sport)
  A validated questionnaire that quantifies quality of life and life satisfaction in pediatric and adolescent populations.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 6-months post initial visit
  A validated questionnaire that quantifies quality of life and life satisfaction in pediatric and adolescent populations.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 12-months post initial visit
  A validated questionnaire that quantifies quality of life and life satisfaction in pediatric and adolescent populations.
Tampa Scale for Kinesiophobia-11 (TSK-11) | Assessed at 1 day initial visit
  Questionnaire designed to assess patient fear of movement.
Tampa Scale for Kinesiophobia-11 (TSK-11) | At follow up visit, up to 3 months post initial visit
  Questionnaire designed to assess patient fear of movement.
Tampa Scale for Kinesiophobia-11 (TSK-11) | 1 day (At clearance visit to return to sport)
  Questionnaire designed to assess patient fear of movement.
Tampa Scale for Kinesiophobia-11 (TSK-11) | 6-months post initial visit
  Questionnaire designed to assess patient fear of movement.
Tampa Scale for Kinesiophobia-11 (TSK-11) | 12-months post initial visit
  Questionnaire designed to assess patient fear of movement.

SECONDARY OUTCOMES:
Injury location and type questionnaire | 1 day Initial visit
  Patient-reported details of their musculoskeletal injury, including injury location and type. Also asks for details regarding the participant's pain rating, duration of pain, and the impact the injury has on sport participation.
Level of Specialization | 1 day (At clearance visit to return to sport)
  Questionnaire designed to identify an athlete's level of sport specialization.
Level of Specialization | 6-months post initial visit
  Questionnaire designed to identify an athlete's level of sport specialization.
Level of Specialization | 12-months post initial visit
  Questionnaire designed to identify an athlete's level of sport specialization.
Injury History | Assessed at the patient's 1 day initial visit.
  Patient-reported history of previous musculoskeletal injuries.
Pittsburgh Sleep Quality Index (PSQI) | Assessed at initial 1 day visit
  Questionnaire used to determine the participant's quality of sleep.
Pittsburgh Sleep Quality Index (PSQI) | At follow up visit, up to 3 months post initial visit
  Questionnaire used to determine the participant's quality of sleep.
Pittsburgh Sleep Quality Index (PSQI) | 1 day (At clearance visit to return to sport)
  Questionnaire used to determine the participant's quality of sleep.
Pittsburgh Sleep Quality Index (PSQI) | 6-months post initial visit
  Questionnaire used to determine the participant's quality of sleep.
Pittsburgh Sleep Quality Index (PSQI) | 12-months post initial visit
  Questionnaire used to determine the participant's quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Sweeney, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hart E, Meehan WP 3rd, Bae DS, d'Hemecourt P, Stracciolini A. The Young Injured Gymnast: A Literature Review and Discussion. Curr Sports Med Rep. 2018 Nov;17(11):366-375. doi: 10.1249/JSR.0000000000000536. PMID 30407945
- [Background] Beleckas CM, Prather H, Guattery J, Wright M, Kelly M, Calfee RP. Anxiety in the orthopedic patient: using PROMIS to assess mental health. Qual Life Res. 2018 Sep;27(9):2275-2282. doi: 10.1007/s11136-018-1867-7. Epub 2018 May 8. PMID 29740783
- [Background] Lim SW, Shiue YL, Ho CH, Yu SC, Kao PH, Wang JJ, Kuo JR. Anxiety and Depression in Patients with Traumatic Spinal Cord Injury: A Nationwide Population-Based Cohort Study. PLoS One. 2017 Jan 12;12(1):e0169623. doi: 10.1371/journal.pone.0169623. eCollection 2017. PMID 28081205
- [Background] Mainwaring LM, Hutchison M, Bisschop SM, Comper P, Richards DW. Emotional response to sport concussion compared to ACL injury. Brain Inj. 2010;24(4):589-97. doi: 10.3109/02699051003610508. PMID 20235761
- [Background] Xanthopoulos MS, Benton T, Lewis J, Case JA, Master CL. Mental Health in the Young Athlete. Curr Psychiatry Rep. 2020 Sep 21;22(11):63. doi: 10.1007/s11920-020-01185-w. PMID 32954448
- [Background] Mauck B, Kelly D, Sheffer B, Rambo A, Calandruccio JH. Gymnast's Wrist (Distal Radial Physeal Stress Syndrome). Orthop Clin North Am. 2020 Oct;51(4):493-497. doi: 10.1016/j.ocl.2020.06.012. Epub 2020 Aug 13. PMID 32950218
- [Background] Putukian M. The psychological response to injury in student athletes: a narrative review with a focus on mental health. Br J Sports Med. 2016 Feb;50(3):145-8. doi: 10.1136/bjsports-2015-095586. Epub 2015 Dec 30. PMID 26719498
- [Background] Pluhar E, McCracken C, Griffith KL, Christino MA, Sugimoto D, Meehan WP 3rd. Team Sport Athletes May Be Less Likely To Suffer Anxiety or Depression than Individual Sport Athletes. J Sports Sci Med. 2019 Aug 1;18(3):490-496. eCollection 2019 Sep. PMID 31427871
- [Background] McGuine TA, Winterstein A, Carr K, Hetzel S, Scott J. Changes in self-reported knee function and health-related quality of life after knee injury in female athletes. Clin J Sport Med. 2012 Jul;22(4):334-40. doi: 10.1097/JSM.0b013e318257a40b. PMID 22627649
- [Background] Valovich McLeod TC, Bay RC, Parsons JT, Sauers EL, Snyder AR. Recent injury and health-related quality of life in adolescent athletes. J Athl Train. 2009 Nov-Dec;44(6):603-10. doi: 10.4085/1062-6050-44.6.603. PMID 19911086
- [Background] Filbay S, Pandya T, Thomas B, McKay C, Adams J, Arden N. Quality of Life and Life Satisfaction in Former Athletes: A Systematic Review and Meta-Analysis. Sports Med. 2019 Nov;49(11):1723-1738. doi: 10.1007/s40279-019-01163-0. PMID 31429036
- [Background] Jayanthi NA, Post EG, Laury TC, Fabricant PD. Health Consequences of Youth Sport Specialization. J Athl Train. 2019 Oct;54(10):1040-1049. doi: 10.4085/1062-6050-380-18. PMID 31633420
- [Background] Pasulka J, Jayanthi N, McCann A, Dugas LR, LaBella C. Specialization patterns across various youth sports and relationship to injury risk. Phys Sportsmed. 2017 Sep;45(3):344-352. doi: 10.1080/00913847.2017.1313077. Epub 2017 Apr 10. PMID 28351225
- [Background] Li H, Moreland JJ, Peek-Asa C, Yang J. Preseason Anxiety and Depressive Symptoms and Prospective Injury Risk in Collegiate Athletes. Am J Sports Med. 2017 Jul;45(9):2148-2155. doi: 10.1177/0363546517702847. Epub 2017 Apr 25. PMID 28441037
- [Background] Chang C, Putukian M, Aerni G, Diamond A, Hong G, Ingram Y, Reardon CL, Wolanin A. Mental health issues and psychological factors in athletes: detection, management, effect on performance and prevention: American Medical Society for Sports Medicine Position Statement-Executive Summary. Br J Sports Med. 2020 Feb;54(4):216-220. doi: 10.1136/bjsports-2019-101583. Epub 2019 Dec 6. PMID 31810972